CLINICAL TRIAL: NCT07204769
Title: Microbiological Characterization and Antibiotic Resistance Profiling of Providencia Spp,: An Emerging Pathogen Isolated From Urinary Tract Infections.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Tareq Diab, Teaching assistant at Medical microbiology and Immunology department, Assiut University
Other Study IDs: Providencia UTI
Record Dates: First submitted 2025-09-22; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Drug Collateral Sensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antibiotic sensitivity — Molecular characterization of multidrug-resistance gene antibiotics.

SUMMARY:
Aims of the Research:

1. Isolation and identification of Providencia spp. from UTIs.
2. Genotypic confirmation of Providencia isolates.
3. Determination of antimicrobial sensitivity patterns of isolated Providencia spp.
4. Characterization of some virulence factors of Providencia spp.
5. Molecular characterization of multidrug-resistance gene antibiotics.
6. Determination of risk factors for Providencia UTIs.

DETAILED DESCRIPTION:
Urinary tract infections (UTIs) are among the most common bacterial infections worldwide, with Escherichia coli, Klebsiella spp., Proteus spp., and Pseudomonas spp. representing the majority of isolated pathogens in both community and hospital settings. Providencia spp., although historically considered uncommon, are increasingly recognized as opportunistic pathogens.

International surveillance studies report that Providencia accounts for ~1-2% of urinary isolates, with higher prevalence (up to 6-12%) in catheter-associated infection.

The Providencia genus, nestled within the Enterobacterales order as part of Proteus and Morganella relatives, consists of Gram-negative bacteria that are adept at producing urease .

The genus includes 14 distinct species, with Providencia rettgeri, Providencia stuartii, Providencia alcalifaciens, and Providencia hangzhouensis standing out due to their pronounced relevance to human infections. Renowned for their association with urinary tract infections, these pathogens also possess the capability to inflict a broader spectrum of severe ailments, such as ocular diseases,peritonitis, neonatal septicemia or bloodstream infections and meningitis.

Providencia stuartii is able to adhere to and invade HeLa-M epithelial cell line.

They form biofilms and have several virulence genes . Providencia spp. may be susceptible to third- and fourth-generation cephalosporins, aztreonam, imipenem, and meropenem. Providencia species have variable susceptibilities to fluoroquinolones, aminoglycosides, and trimethoprim- sulfamethoxazole (TMP-SMX). Generally, Providencia spp. are frequently resistant to tetracyclines, penicillins, and first- and second- generation cephalosporins .

Providencia spp.are intrinsically resistant to polymyxins and tigecycline, which are considered last- resort antibiotics for other resistant pathogens .

In Egypt, several studies have investigated the prevalence of UTI pathogens, consistently reporting E. coli, Klebsiella spp., and Proteus spp. as the most frequent isolates .

However, no published Egyptian data specifically describe the prevalence, antimicrobial resistance patterns, or clinical significance of Providencia spp. in UTIs.

This gap highlights the need for focused research on Providencia in the Egyptian context. Studying its frequency, antibiotic resistance mechanisms, and clinical relevance would not only provide novel insights but also contribute to improving diagnosis, empirical therapy, and infection control strategies in Egyptian hospitals .

ELIGIBILITY:
Inclusion Criteria:

Patients with UTI diagnosed through clinical examination and urine analysis. Informed consent will be obtained from each patient before Participation in the study.

Exclusion Criteria:

1. Patients currently on antibiotics.
2. Patients with any anatomical abnormalities in the urinary tract C) Patients having UTI by gram +ve organisms.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with UTI diagnosed through clinical examination and urine analysis.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Determination of prevalence of Providencia species refers specifically to urinary tract infection patients with gram-negative bacterial isolates. | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aya Tareq Diab, Bachelor's degree, Principal Investigator — Assiut University; Prof: Mona Hussein Abdel-Rahim, PhD, Study Director — Assiut University; Dr. Rawhia Fathy Abdel Hamid, Doctorate, Study Chair — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Çetin ET, et al. Providencia spp. in nosocomial urinary infections. Turk J Med Sci. 1998;28(1):59-62
- [Background] Ewing WH. The tribe Proteeae: its nomenclature and taxonomy. Int J Syst Evol Microbiol. 1962;12(3):93-102
- [Background] Charbek EPN. Providencia infections treatment & management: medical care, surgical care, consultations. Medscape. 2019
- [Background] Rose WE, Rybak MJ. Tigecycline: first of a new class of antimicrobial agents. Pharmacotherapy. 2006 Aug;26(8):1099-110. doi: 10.1592/phco.26.8.1099. PMID 16863487
- [Background] Guidone GHM, Cardozo JG, Silva LC, Sanches MS, Galhardi LCF, Kobayashi RKT, Vespero EC, Rocha SPD. Epidemiology and characterization of Providencia stuartii isolated from hospitalized patients in southern Brazil: a possible emerging pathogen. Access Microbiol. 2023 Oct 18;5(10):000652.v4. doi: 10.1099/acmi.0.000652.v4. eCollection 2023. PMID 37970084
- [Background] Kurmasheva N, Vorobiev V, Sharipova M, Efremova T, Mardanova A. The Potential Virulence Factors of Providencia stuartii: Motility, Adherence, and Invasion. Biomed Res Int. 2018 Feb 21;2018:3589135. doi: 10.1155/2018/3589135. eCollection 2018. PMID 29682537
- [Background] Dong X, Xiang Y, Yang P, Wang S, Yan W, Yuan Y, Zhou S, Zhou K, Liu J, Zhang Y. Novel Providencia xianensis sp. nov.: A multidrug-resistant species identified in clinical infections. Eur J Clin Microbiol Infect Dis. 2024 Jul;43(7):1461-1467. doi: 10.1007/s10096-024-04821-y. Epub 2024 May 7. PMID 38714595
- [Background] O'Hara CM, Brenner FW, Miller JM. Classification, identification, and clinical significance of Proteus, Providencia, and Morganella. Clin Microbiol Rev. 2000 Oct;13(4):534-46. doi: 10.1128/CMR.13.4.534. PMID 11023955
- [Background] Wie SH. Clinical significance of Providencia bacteremia or bacteriuria. Korean J Intern Med. 2015 Mar;30(2):167-9. doi: 10.3904/kjim.2015.30.2.167. Epub 2015 Feb 27. No abstract available. PMID 25750557